CLINICAL TRIAL: NCT02873533
Title: Pilot Project - Prospective Longitudinal Cohort of Patients Over 70 Years With Malignant Solid Tumors: Modification of Quality of Life Based on Objective Geriatric Tests
Brief Title: Modification of the Quality of Life Based on Objective Geriatric Tests
Acronym: MEGERIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011/11 MEGERIA; 2012-A01168-35 (Other: ANSM ID RCB)
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Elderly Patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A-Elderly patients with cancer (Other): geriatric care and longitudinal follow up
  Interventions: Other: geriatric care and longitudinal follow up

INTERVENTIONS:
Other: geriatric care and longitudinal follow up — geriatric care and longitudinal follow up

SUMMARY:
The analysis of this study will achieve an improvement in the management of patients over 70 years with adaptation of chemotherapy regimens after analysis of the subject and its psychosocial environment.

The analysis of socio-economic impacts will implement actions to optimize the care of the elderly while emphasizing the value of management / cost of care.

DETAILED DESCRIPTION:
Quality of life is defined as "an individual's perception of his place in life, in the context of culture and value system in which he lives, in relation to its goals, expectations, standards and concerns "(WHO 1993).

This concept refers to multiple dimensions, both objective and subjective:

* The physical condition of the person, his functional abilities;
* His somatic sensations;
* His psychological health;
* His social status, relational environment.

This concept focuses on perception's basics. Quality of life is a criteria supposed to be objective even though it is subject to subjective interpretation at the highest point. Indeed, if the quality of life varies depending on the discretion of each person, it also changes over time: it refers to a situation at a given moment and not to a stable state.

Therefore in this study, it seemed appropriate to show the concept of "quality of life objective" which is linked to objective data measures recognized criteria for evaluating the elderly. These criteria are repeatable, validated and not dependent operator.

This process completely matches with the actions promoted by the 2009-2013 Cancer Plan (measures 23 and 26) on the basis of an improvement of:

* The quality of consideration of the psychosocial dimension (customization accompaniment, living environment, social, involvement, ..)
* The quality of the integration of physical and psychological dangers inherent to this weakness situation induced by cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 70 years,
* Patient with a solid malignant tumor,
* Patients for whom a first line chemotherapy is theoretically indicated
* Patient chemotherapy naive,
* Performance Index (PS) <4

Exclusion Criteria:

* Patient not understanding or do not speak French,
* Patients with any severe psychopathological disorder preventing the completion of the questionnaire or invalidating a priori measures of the questionnaire

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-03; Primary Completion 2019-03 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Measuring quality of life according to geriatric questionnaires | 36 months
  Activities of Daily Living Questionnaire

SECONDARY OUTCOMES:
Geriatric Screening Test fragilities and comorbidities | 36 months
  Mini Mental State Examination

CONTACTS AND LOCATIONS:
Overall Officials: Véronique MARI, md, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided